CLINICAL TRIAL: NCT05378815
Title: Platelet-rich Plasma in Symptomatic Knee Osteoarthritis: a Randomized, Double-blind, Placebo-controlled, Multicentre Trial
Brief Title: Platelet-rich Plasma in Symptomatic Knee Osteoarthritis
Acronym: PIKOA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP200819; 2021-A00742-39 (Other: N° IDRCB)
Record Dates: First submitted 2022-05-09; First posted 2022-05-18 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Platelet rich plasma; PRP; Placebo controlled trial
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Randomised, double blinded, placebo-controlled trial comparing 3 intra-articular injections of PRP (Regenkit) and NaCl in patients with symptomatic knee osteoarthritis
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In this trial, the patient, the investigator performing the intra-articular injection and the investigator assessing the outcomes will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRP group (Experimental): PRP will be prepared with A-CP-T-20 kit provided by the RegenLab laboratory. This is a 2B medical device with the CE mark. 5mL will be injected in knee under ultrasound guidance.
  The PRP extracted using this kit is poor in leukocytes, has a platelet concentration multiplied by 1.6 on average compared to circulating blood and is not activated (P2Bbeta according to the PAW classification; 3B according to the Mishra's classification).
  Interventions: Procedure: PRP injection
- Placebo group (Placebo Comparator): 5 mL of NaCl will be injected in knee under ultrasound guidance.
  Interventions: Procedure: Placebo injection

INTERVENTIONS:
Procedure: PRP injection — 3 weekly intra-articular injections of 5mL PRP under ultrasound guidance
  Arms: PRP group
Procedure: Placebo injection — 3 weekly intra-articular injections of 5mL NaCL under ultrasound guidance
  Arms: Placebo group

SUMMARY:
Intro:

Platelet rich plasma (PRP) is largely used in various musculoskeletal disorders such as chronic tendinopathies but also osteoarthritis (OA). Several therapeutic trials evaluating the effectiveness of intra-articular PRP injections in knee OA as well as meta-analyses have already been published. Most of them have compared PRP to Hyaluronic Acid (HA). Their design was very heterogeneous in terms of PRP characteristics and injection protocol. Moreover, the number of patients included was often very low. Only few studies have compared PRP to placebo (physiological serum) and presented the same methodological limitations (limited number of patients, heterogeneous protocols in terms of number and frequency of injections, characteristics of PRP, etc.).

Given the insufficient level of evidence related to these limitations, PRP injections are not recommended in the treatment of symptomatic knee OA by the main scientific societies such as American College of Rheumatology (ACR), Osteoarthritis Research Society International (OARSI), American Academy of Orthopedic Surgeons (AAOS) and French Society of Rheumatology (SFR). Experts in the field agree on the need for a placebo-controlled trial with hihg methodological quality and simple design in order to conclude with a good level of evidence to the benefit or not of this new therapeutic weapon in symptomatic knee osteoarthritis of moderate radiographic severity.

DETAILED DESCRIPTION:
Hypothesis/Objective:

The main objective of this trial is to assess the pain decrease over the last 48 hours assessed by simple numerical scale (NRS) at W14 after 3 weekly injections of PRP (W0, W1 and W2) compared to 3 injections of an equivalent volume of physiological serum in patients suffering from a knee osteoarthritis of moderate radiological severity [Kellgren and Lawrence (KL) 2 or 3].

The secondary objectives will aim to compare the decrease in the level of pain and functional assessed by NRS at W8 and W26, WOMAC scores at W8, W14 and W26, by OMERACT-OARSI response at W8, W14 and W26, in EQ5D-5L score at W8, W14 and W26 between PRN and placebo group. We will also assess the decrease in the consumption of analgesics at W8, W14 and W26 and the decrease in serum level of Coll2-1, Coll2-1 NO₂ and increase in PIIANP level at W8 and W14

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 79
* Symptomatic knee OA according to ACR criteria evolving for more than 3 months
* Predominantly femoro-tibial pain
* KL 2 or 3 on femorotibial compartment on X-rays of less than 6 months
* ENS ≥ 40/100 (with or without usual analgesic treatments)
* Failures or contraindications to conventional treatments (analgesics, NSAIDs)
* Patient able to understand the requirements of the trial and having signed a free and informed consent before entering the study
* Patient able to read and understand written instructions
* Patient able to complete the self-questionnaires
* Use of effective contraception in premenopausal women

Exclusion Criteria:

* Other pathologies of the lower limbs interfering with the evaluation of knee osteoarthritis (symptomatic hip OA, Lumbar pain…)
* Symptomatic contralateral knee OA with NRS ≥ 40/100
* Predominant patellofemoral symptoms
* Radiographic knee OA stage 1 or 4 of KL
* Predominant radiographic patellofemoral OA
* History of target knee surgery with material
* History of inflammatory or microcrystalline rheumatism
* History of fibromyalgia
* Morbid obesity (BMI> 40kgs / m2)
* Inflammatory flare (KOFUS score ≥ 7)
* Use of opioids in the month prior to inclusion
* Patient refusing to stop NSAIDs during the study and conventional analgesics 48 hours
* History of infection of the target knee
* Presence of chondrocalcinosis on the frontal x-ray
* Previous PRP injection
* Injection of HA or CS into the target knee during the last 3 months
* History of hemostasis disorders or taking a curative dose of anticoagulant
* Treatment with antiplatelet agents [Acetylsalicylic acid (Aspegic, Kardegic, Duoplavin, Resitune, Asasantine), Clopidogrel (Plavix, Duoplavin), Dipyridamole (Persantine, Cleridium, Asasantine)]
* Haematological disease in progress or in remission for less than 5 years (malignant hemopathies, myelodysplasia, autoimmune thrombocytopenia)
* Thrombocytopenia (<150,000 platelets)
* Patient undergoing treatment with chemotherapy or immunosuppressive drugs
* Infection at the time of inclusion (bacterial infection and / or presence of fever and / or taking antibiotics)
* Participation in a clinical trial on knee osteoarthritis during the last year
* Participation in any clinical trial completed less than 3 months ago
* Patient whose mental state does not allow him to understand the nature, objectives and possible consequences of the study
* Patient under legal protection (curatorship or guardianship)
* Pregnant woman or planning to become pregnant during the study or breastfeeding

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in global pain intensity in the target knee over the past 48 hours as assessed by Numeric Rating Scale (NRS) between week 0 and week 14 | between week 0 and week 14

SECONDARY OUTCOMES:
Intensity of global pain in the target knee over the last 48 hours evaluated by NRS between week 0 and week 26 | between week 0 and week 26
WOMAC score | between week 0 and week 26
  The WOMAC score is a composite score widely used in international studies on knee osteoarthritis. This is a self-administered questionnaire comprising 3 sub-scores assessing pain (5 items), function (17 items) and stiffness (2 items). Each item is measured on a graduated scale from 0 to 100 (100 corresponding to the most severe symptoms). An average out of 100 will be calculated for each sub score and then for the total WOMAC score. The WOMAC score will be calculated before the first injection (W0) and at W8 and W14.
OMERACT-OARSI response | between week 0 and week 26
  The OMERACT-OARSI response was developed by international scientific societies working on osteoarthritis in order to identify patients with a significant and clinically relevant response to a therapeutic strategy or to a given treatment. It is defined as either an improvement in the WOMAC pain score or the WOMAC score based on at least 50% and at least 20 points out of 100, or an improvement of at least 20% and at least 10 points out of 100 for 2 of the 3 following criteria: WOMAC pain score, WOMAC function score and overall assessment of symptoms by the patient (measured by graduated scale from 0 to 100). This response will be evaluated at W8 and W14.
EQ5D-5L score | between week 0 and week 26
  The EQ5D-5L score is a composite quality of life score assessing 5 different areas (mobility, personal care, daily activities, pain, anxiety) and validated in osteoarthritis and chronic pain. Each item is measured on a scale of 1 (most favorable condition) to 5 (most unfavorable condition) depending on the severity of symptoms. The EQ5D-5L score will be calculated before the first injection (W0), at W8 and at W14.
Number of level 1 or 2 analgesics consumed | between week 0 and week 26
  The consumption of analgesics will be evaluated at WO, W8, W14 and W26. The number and dose of level 1 or 2 analgesics consumed during the week preceding the visit will be noted (D-7 to D-2 before each assessment, patients not being authorized to take analgesics within 48 hours before the assessment). A notebook will be given to the patient so that he notes each analgesic taken with dosage and daily frequency.
drug dose of level 1 or 2 analgesics consumed | between week 0 and week 26
  The consumption of analgesics will be evaluated at WO, W8, W14 and W26. The number and dose of level 1 or 2 analgesics consumed during the week preceding the visit will be noted (D-7 to D-2 before each assessment, patients not being authorized to take analgesics within 48 hours before the assessment). A notebook will be given to the patient so that he notes each analgesic taken with dosage and daily frequency.
Collection of adverse events | between week 0 and week 26
Serum biomarker assay Coll2-1 | between week 0 and week 14
Serum biomarker assay Coll2-1 NO₂ | between week 0 and week 14
Serum biomarker assay PIIANP | between week 0 and week 14

CONTACTS AND LOCATIONS:
Overall Officials: Florent Eymard, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Henri Mondor, Créteil, Val-De-Marne
  - Florent Eymard, Créteil

REFERENCES:
- [Derived] Eymard F, Oubaya N, Ornetti P, Sellam J, Richette P, Chevalier X; PIKOA study group. Protocol for a multicentre randomised triple-blind controlled trial assessing the clinical efficacy of intra-articular platelet-rich plasma injections versus placebo in symptomatic knee osteoarthritis (PIKOA). BMJ Open. 2024 Nov 29;14(11):e085025. doi: 10.1136/bmjopen-2024-085025. PMID 39615889